CLINICAL TRIAL: NCT01550627
Title: Study of Possible Effects of Intravenous Fluid Supplementation on Serum Bilirubin Levels and Cardiorespiratory Parameters in Preterm Infants During Phototherapy
Brief Title: Effect of Intravenous Fluid Supplementation on Serum Bilirubin and Cardiorespiratory Parameters in Preterm Infants During Phototherapy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, Stefanie Junge, (MD), University of Jena
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2127-10/09
Record Dates: First submitted 2012-02-07; First posted 2012-03-12 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2012-03

CONDITIONS: Hyperbilirubinemia
Keywords: preterm infants < 32 weeks of gestation
MeSH Terms: conditions — Hyperbilirubinemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- extra-fluid (Active Comparator): The study group received an extra intravenous fluid intake of 20% of the total fluid demand per 24 hours of NaCl 0,9% during each two hour period of phototherapy (12h total per day).
  Interventions: Other: extra fluid/iv fluid supplementation during phototherapy
- non extra fluid (control group) (Placebo Comparator): The control group received the previous fluid regime, as intravenous fluid was given constantly, without a specific guideline according to extra fluid intake.
  Interventions: Other: Non extra fluid

INTERVENTIONS:
Other: extra fluid/iv fluid supplementation during phototherapy — The study group received an extra intravenous fluid intake of 20% of the total fluid demand per 24 hours of NaCl 0,9% during each two hour period of phototherapy (12h total per day). The extra fluid intake was interrupted during the 12 hours break of phototherapy.
  Arms: extra-fluid
Other: Non extra fluid — Control placebo The control group received the previous fluid regime, as intravenous fluid was given constantly, without a specific guideline according to extra fluid intake.
  Arms: non extra fluid (control group)

SUMMARY:
The aim of the study was to evaluate the influence of a systematic extra intravenous fluid supplementation during phototherapy in comparison to a fluid supplementation due to short term demand in preterm infants.

DETAILED DESCRIPTION:
60 preterm infants (GA ≤ 32 week) were assigned randomly to either receive a fluid supplementation due to short term demand (control group, n=30;) or a 20% extra fluid supplementation (study group, n=30) during intermediate phototherapy.

Collected data:

* cardiorespiratory parameters(heart rate, blood pressure, SaO2 and capillary refill time, breathing rate, temperature) and a pain score was completed at the first day of phototherapy
* The maximum total serum bilirubin levels (TSB) within one week after onset of phototherapy

ELIGIBILITY:
Inclusion Criteria:

* Hyperbilirubinemia

Exclusion Criteria:

* Preterm infants > 33 weeks of gestation

Ages: 1 Week to 1 Week | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2007-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The maximum total serum bilirubin levels | within one week after onset of phototherapy
  The maximum total serum bilirubin levels within on week after onset of phototherapy

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Jena, Jena, Jena, Germany